CLINICAL TRIAL: NCT01594255
Title: A Randomized, Partially Blinded, 4-period, Crossover Study to Assess the Effects of Single-dose AEB071 Administration (300 and 900 mg) on Electrocardiographic QT Intervals Compared to Placebo in Healthy Volunteers
Brief Title: CAEB071 Thorough QTc Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CAEB071A2115
Record Dates: First submitted 2012-05-03; First posted 2012-05-09 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Healthy volunteer; QT intervals; ECG; QT/QTc interval prolongation and proarrhythmic potential for non-antiarrhythmic drugs
MeSH Terms: interventions — sotrastaurin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- AEB071 300 mg (Experimental)
  Interventions: Drug: sotrastaurin
- AEB071 900 mg (Experimental)
  Interventions: Drug: sotrastaurin
- Placebo to AEB071 (Placebo Comparator)
  Interventions: Drug: placebo to sotrastaurin
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Avelox

INTERVENTIONS:
Drug: sotrastaurin
  Arms: AEB071 300 mg
Drug: sotrastaurin
  Arms: AEB071 900 mg
Drug: placebo to sotrastaurin
  Arms: Placebo to AEB071
Drug: Avelox
  Arms: Moxifloxacin

SUMMARY:
This study has been designed in compliance with the ICH-E14 guideline 2005 to evaluate the QT/QTc interval prolongation and proarrhythmic potential for non-antiarrhythmic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects age 18 to 50 years (including both) of age included, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.

Exclusion Criteria:

* Smokers and tobacco product users (in the previous 3 months).
* Use of any prescription drugs, herbal supplements, within four (4) weeks prior to initial dosing, and/or over-the-counter (OTC) medication, dietary supplements (vitamins included) within two (2) weeks prior to initial dosing.
* A marked baseline prolongation of QT/QTcF interval
* Presence of clinically significant illness
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change in the corrected QT interval (QTc) in healthy volunteers as compared to placebo. | 24 hours

SECONDARY OUTCOMES:
Change in concentration of exposure-response AEB071 and AEE800 (a metabolite of AEB071) concentrations compared to cardiac repolarization intervals | 24 hours
Tolerability of 300 and 900 mg of AEB071. | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigational Site, Austin, Texas, United States